CLINICAL TRIAL: NCT00436046
Title: Type 1 Interferon as a Mucosal Adjuvant for Influenza Vaccine Given Intranasally
Brief Title: Interferon as a Mucosal Adjuvant for Influenza Vaccine Given Intranasally
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Director, ORA, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06-0074; N01AI30039C; N01AI30039 (NIH)
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Results first posted 2008-11-18 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2009-10

CONDITIONS: Influenza
Keywords: interferon, vaccine, influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Group 1: 0.6 ml of IVV (Active Comparator): 30 subjects to receive 0.6 ml of inactivated influenza virus vaccine (IVV).
  Interventions: Biological: Trivalent inactivated influenza virus vaccine (2006-2007 formulation)
- Group 3: 0.7 ml of IVV + 10M units of IFN (Experimental): 30 subjects to receive 0.7 ml of IVV containing 10M units of interferon (IFN).
  Interventions: Biological: Trivalent inactivated influenza virus vaccine (2006-2007 formulation); Biological: Type 1 interferon
- Group 2: 0.6 ml of IVV + 1M unit of IFN (Experimental): 30 subjects to receive 0.6 ml of IVV containing 1M units of interferon (IFN).
  Interventions: Biological: Trivalent inactivated influenza virus vaccine (2006-2007 formulation); Biological: Type 1 interferon

INTERVENTIONS:
Biological: Trivalent inactivated influenza virus vaccine (2006-2007 formulation) — Commercially available trivalent inactivated influenza virus vaccine without or with 1 of 2 dosages of commercially available type 1 interferon administered once by nasal instillation. Dosages: 0.6 ml of IVV or 0.7 ml of IVV.
Biological: Type 1 interferon — Commercially available lyophilized IFN; dosages 1 M unit (Mu) of IFN; 10 M units (Mu) of IFN.
  Arms: Group 2: 0.6 ml of IVV + 1M unit of IFN; Group 3: 0.7 ml of IVV + 10M units of IFN

SUMMARY:
Influenza is a virus infection that causes sickness from the nose to the lungs. It is thought that type 1 interferon (a protein that helps the immune system fight viruses) will make flu vaccines more effective. This study will determine if type 1 interferon added to a specific flu vaccine will help the immune system of healthy adults fight off infection better than vaccine alone. Ninety volunteers, ages 18-40, will participate in this study. They will attend 3 study visits and have a final follow-up study visit, email, or phone call about six months after the vaccination. Volunteers will receive a single dose of study vaccine sprayed into the nose. Study procedures including blood samples and nasal washes (the inside of the nose is washed out) will be collected to evaluate immune system responses.

DETAILED DESCRIPTION:
Influenza is primarily a virus infection of the respiratory tract mucosa from the nose to the terminal bronchioles. Immunity to influenza virus infection is mediated primarily by antibody in respiratory secretions at the mucosal surface. To meet the need for improved inactivated vaccines, one potential approach is to increase the frequency and magnitude of antibody in secretions by administering inactivated influenza virus vaccine (IVV) intranasally and to optimize responses by including a mucosal adjuvant. The primary hypothesis of this study is that Type 1 interferon (IFN) will provide an adjuvant effect at the respiratory mucosal surface for production of IgA and/or IgG antibody to the influenza strains when added to IVV and administered intranasally. The primary objective of the study is to determine whether including type 1 IFN with IVV, administered intranasally, to healthy adults will enhance antibody responses in nasal secretions compared to intranasal administration of IVV alone. This is a single-center, randomized, double-blind, clinical trial to determine if type 1 IFN will act as a mucosal adjuvant for antibody responses to influenza viruses after administration with IVV intranasally. Subjects will be healthy adults between the ages of 18 and 40. The study will enroll 30 subjects in each of three groups, a group given 0.6 ml of IVV, a group given 0.6 ml of IVV containing 1M units of IFN and a group given 0.7 ml of IVV containing 10M units of IFN. The vaccine or vaccine/interferon combination will be administered to the subjects intranasally once. Blood and nasal secretions will be obtained before vaccination and again two and four weeks after immunization. Each subject will be asked to complete a memory aid for seven days and to report any unexpected adverse events (AEs) to study personnel. The subject will report to the clinic or be contacted by phone or e-mail at six months after vaccination regarding occurrence of any unreported serious adverse events (SAEs). The three nasal secretions will be used for testing for IgA and IgG antibody to the A/H1N1 and A/H3N2 HA in enzyme-linked immunosorbent assay (ELISA) tests. The three blood samples will be tested in HAI and neutralization tests for antibody to the A/H1N1 and A/H3N2 vaccine antigens.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female (as indicated by a negative urine pregnancy test immediately prior to vaccine administration) between the ages of 18 and 40 years.
* Women of childbearing potential who are at risk of becoming pregnant must agree to practice adequate contraception (e.g., barrier method, abstinence, and licensed hormonal methods) for at least 3 months after immunization.
* Is in good health, as determined by vital signs (heart rate, blood pressure, oral temperature), medical history and a targeted physical examination based on medical history.
* Able to understand and comply with planned study procedures.
* Provides informed consent prior to any study procedures and is available for all study visits.

Exclusion Criteria:

* Has a known allergy to eggs, chicken protein or other components of the vaccine.
* Has a positive urine pregnancy test prior to vaccination (if female of childbearing potential), is lactating, or has the intention to become pregnant within 3 months of receipt of vaccine.
* Is undergoing immunosuppression as a result of an underlying illness or treatment.
* Has an active neoplastic disease or a history of any hematologic malignancy.
* Is using oral or parenteral steroids or other immunosuppressive or cytotoxic drugs.
* Has used any nasal or aerosol treatments in the past 2 weeks or likely to use any in the next 2 weeks.
* Has a diagnosis of hay fever or asthma.
* Has a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* Has a diagnosis of schizophrenia, bipolar disease or other major psychiatric diagnosis.
* Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
* Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (this includes, but is not limited to: known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients).
* Has a history of severe reactions following immunization with contemporary influenza virus vaccines.
* Has an acute illness, including an oral temperature greater than 100.4 degrees F, within 1 week prior to vaccination.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in the study, or expects to receive an experimental agent during the 6-month study period.
* Is planning to enroll in another clinical trial at any time during the study period.
* Has known active human immunodeficiency virus, hepatitis B or hepatitis C infection.
* Has a history of alcohol or drug abuse in the last 5 years.
* Has a history of Guillain-Barre syndrome.
* Has received the 2006-2007 formulation influenza vaccine by injection or by nose drops (fall of 2006 or since).
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2007-03; Primary Completion 2007-04 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy ambulatory adults were recruited from the surrounding community of the research clinic from March 16, 2007 through March 21, 2007.
Groups:
- IVV With 1M IFN: IVV (inactivated influenza virus vaccine) plus 1 Molar unit of IFN (Interferon): 0.6ml of the mixture will be given [0.5 ml of vaccine plus 0.1 ml (1 Molar unit) of IFN].
- IVV Without IFN: IVV only: 0.6 ml of IVV alone (0.5 ml of vaccine plus 0.1 ml of saline).
- IVV With 10M IFN: IVV plus 10 Molar units of IFN: 0.7 ml of the mixture will be given [0.5 ml of vaccine plus 0.2 ml (10 Molar units) of IFN].
Period: Overall Study
Arm/Group | IVV With 1M IFN | IVV Without IFN | IVV With 10M IFN
Started | 32 | 32 | 31
Completed | 32 | 32 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVV With 1M IFN | IVV Without IFN | IVV With 10M IFN | Total
Number analyzed (Participants) | 32 | 32 | 31 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 32 | 31 | 31 | 94
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.3 (5.2) | 25.2 (4.8) | 24.7 (4.9) | 25.1 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 23 | 63
  Male | 10 | 14 | 8 | 32
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 31 | 95

OUTCOME MEASURES:

1. Primary Outcome: Antibody Responses in Nasal Secretions to Influenza A/H1N1 and A/H3N2 at 14 Days After Intranasal Immunization.
Description: Number of subjects (frequency) responding with a four-fold or greater increase (magnitude) in titer at day 14 after immunization, relative to pre-immunization levels
Time Frame: 14 days after immunization.
Measure: Number; unit: Participants
Arm/Group | IVV With 1M IFN | IVV Without IFN | IVV With 10M IFN
Number analyzed (Participants) | 32 | 32 | 31
Participants
  IgG to A/New Caledonia/20/99 at Day 14 | 3 | 3 | 5
  IgA to A/New Caledonia/20/99 at Day 14 | 0 | 2 | 1
  IgG to A/Wisconsin/67/2005 at Day 14 | 2 | 3 | 4
  IgA to A/Wisconsin/67/2005 at Day 14 | 3 | 1 | 6

2. Secondary Outcome: Local and/or Systemic Solicited Symptoms After Intranasal Immunization.
Description: Number of participants (frequency) reporting solicited (systematically collected on a Memory Aid) reactogenicity events of any severity and number reporting severe occurrences.
Time Frame: 0-7 days following immunization
Measure: Number; unit: Participants
Arm/Group | IVV With 1M IFN | IVV Without IFN | IVV With 10M IFN
Number analyzed (Participants) | 32 | 32 | 31
Participants
  Elevated Oral Temperature - Any severity | 0 | 1 | 0
  Elevated Oral Temperature - Severe | 0 | 0 | 0
  Feverishness - Any severity | 0 | 1 | 2
  Feverishness - Severe | 0 | 1 | 0
  Malaise - Any severity | 7 | 11 | 9
  Malaise - Severe | 0 | 1 | 2
  Myalgia - Any severity | 7 | 5 | 5
  Myalgia - Severe | 0 | 1 | 0
  Headache - Any severity | 14 | 17 | 12
  Headache - Severe | 0 | 0 | 1
  Nausea - Any severity | 1 | 1 | 6
  Nausea - Severe | 0 | 1 | 0
  Nasal Obstruction - Any severity | 9 | 10 | 9
  Nasal Obstruction - Severe | 0 | 0 | 0
  Nasal Discharge - Any severity | 14 | 14 | 10
  Nasal Discharge - Severe | 0 | 0 | 0
  Sneezing - Any severity | 10 | 13 | 9
  Sneezing - Severe | 0 | 0 | 0
  Sore Throat - Any severity | 10 | 10 | 11
  Sore Throat - Severe | 0 | 0 | 0
  Cough - Any severity | 5 | 5 | 8
  Cough - Severe | 0 | 0 | 0
  Any systemic symptom of any severity | 21 | 21 | 20
  Severe systemic symptom | 0 | 1 | 2
  Any local symptom of any severity | 22 | 24 | 20
  Severe local symptom | 0 | 0 | 0
  Any symptom of any severity | 27 | 28 | 26
  Severe symptom | 0 | 1 | 2

3. Secondary Outcome: Serum Antibody Responses (Hemagglutination Inhibition (HAI) and Neutralization) to Influenza A/H1N1 and A/H3N2 at 14 Days After Intranasal Immunization.
Description: Number of subjects (frequency) responding with a four-fold or greater increase (magnitude) in titer at 14 days after immunization, relative to pre-immunization levels.
Time Frame: 14 days after immunization.
Measure: Number; unit: Participants
Arm/Group | IVV With 1M IFN | IVV Without IFN | IVV With 10M IFN
Number analyzed (Participants) | 32 | 32 | 31
Participants
  HAI - A/New Caledonia/20/99 at Day 14 | 13 | 16 | 11
  HAI - A/Wisconsin/67/2005 at Day 14 | 12 | 21 | 7
  Neutralization - A/New Caledonia/20/99 at Day 14 | 12 | 13 | 9
  Neutralization - A/Wisconsin/67/2005 at Day 14 | 13 | 16 | 10

4. Secondary Outcome: Unsolicited Adverse Events After Intranasal Immunization
Description: Number of subjects (frequency) with spontaneous reports of Adverse Events of any severity and severe or higher severity, during the 28 days after vaccination regardless of relatedness. Events reported by more than 5.6% of subjects in any group are reported by MedDRA Preferred Term.
Time Frame: Non-serious AEs are collected through 28 days after vaccination. Serious AEs are collected through 180 days after vaccination.
Population: A reporting threshold of 5.6% was selected after reviewing adverse event rates in healthy adult volunteers in similar studies sponsored by NIAID. We determined 5.6% to be the upper bound of the confidence interval to exclude reporting events that occur in 75% of healthy adults.
Measure: Number; unit: Participants
Arm/Group | IVV With 1M IFN | IVV Without IFN | IVV With 10M IFN
Number analyzed (Participants) | 32 | 32 | 31
Participants
  Abdominal pain upper - Any severity | 2 | 0 | 0
  Abdominal pain upper - Severe | 0 | 0 | 0
  Upper respiratory tract infection - Any severity | 4 | 3 | 3
  Upper respiratory tract infection - Severe | 0 | 1 | 0
  Dysgeusia - Any severity | 2 | 1 | 0
  Dysgeusia - Severe | 0 | 0 | 0
  Pharyngolaryngeal pain - Any severity | 1 | 2 | 1
  Pharyngolaryngeal pain - Severe | 0 | 0 | 0
  Rhinorrhoea - Any severity | 3 | 0 | 1
  Rhinorrhoea - Severe | 0 | 0 | 0
  Dizziness - Any severity | 2 | 0 | 0
  Dizziness - Severe | 0 | 0 | 0
  Dysphonia - Any severity | 0 | 0 | 2
  Dysphonia - Severe | 0 | 0 | 0
  Postnasal drip - Any severity | 0 | 0 | 2
  Postnasal drip - Severe | 0 | 0 | 0
  Diarrhoea - Any severity | 0 | 3 | 0
  Diarrhoea - Severe | 0 | 0 | 0

5. Other Pre Specified Outcome: Serum Antibody Responses (Hemagglutination Inhibition (HAI) and Neutralization) to Influenza B at 14 Days After Intranasal Immunization.
Description: as for outcome 3
Time Frame: 14 days after immunization
Measure: Number; unit: Participants
Arm/Group | IVV With 1M IFN | IVV Without IFN | IVV With 10M IFN
Number analyzed (Participants) | 32 | 32 | 31
Participants
  HAI - B/Malaysia/2506/2004 at Day 14 | 11 | 13 | 8
  Neutralization - B/Malaysia/2506/2004 at Day 14 | 9 | 12 | 8

6. Primary Outcome: Antibody Responses in Nasal Secretions to Influenza A/H1N1 and A/H3N2 at 28 Days After Intranasal Immunization
Description: Number of subjects (frequency) responding with a four-fold or greater increase (magnitude) in titer at day 28 after immunization, relative to pre-immunization levels.
Time Frame: 28 days after immunization.
Measure: Number; unit: Participants
Arm/Group | IVV With 1M IFN | IVV Without IFN | IVV With 10M IFN
Number analyzed (Participants) | 32 | 32 | 31
Participants
  IgG to A/New Caledonia/20/99 at Day 28 | 1 | 3 | 3
  IgA to A/New Caledonia/20/99 at Day 28 | 1 | 3 | 1
  IgG to A/Wisconsin/67/2005 at Day 28 | 3 | 4 | 6
  IgA to A/Wisconsin/67/2005 at Day 28 | 3 | 3 | 4

7. Secondary Outcome: Serum Antibody Responses (Hemagglutination Inhibition (HAI) and Neutralization) to Influenza A/H1N1 and A/H3N2 at 28 Days After Intranasal Immunization.
Description: Number of subjects (frequency) responding with a four-fold or greater increase (magnitude) in titer at 28 days after immunization, relative to pre-immunization levels.
Time Frame: 28 days after immunization
Measure: Number; unit: Participants
Arm/Group | IVV With 1M IFN | IVV Without IFN | IVV With 10M IFN
Number analyzed (Participants) | 32 | 32 | 31
Participants
  HAI - A/New Caledonia/20/99 at Day 28 | 14 | 17 | 11
  HAI - A/Wisconsin/67/2005 at Day 28 | 20 | 23 | 7
  Neutralization - A/New Caledonia/20/99 at Day 28 | 15 | 17 | 10
  Neutralization - A/Wisconsin/67/2005 at Day 28 | 13 | 17 | 8

8. Other Pre Specified Outcome: Serum Antibody Responses (Hemagglutination Inhibition (HAI) and Neutralization) to Influenza B at 28 Days After Intranasal Immunization.
Description: as for outcome 7
Time Frame: 28 days after immunization
Measure: Number; unit: Participants
Arm/Group | IVV With 1M IFN | IVV Without IFN | IVV With 10M IFN
Number analyzed (Participants) | 32 | 32 | 31
Participants
  HAI - B/Malaysia/2506/2004 at Day 28 | 16 | 14 | 9
  Neutralization - B/Malaysia/2506/2004 at Day 28 | 13 | 16 | 13

ADVERSE EVENTS:
Time Frame: Subjects recorded solicited symptoms on a memory aid for 8 days (Day 0-7)following vaccination. Unsolicited non-serious adverse events were collected for 28 days after vaccination and serious adverse events were collected through Day 180
Description: The occurrence of a solicited symptom on any day(s) at any severity within the 8 day (Day 0-7) period was considered one event.
Arm/Group | IVV With 1M IFN | IVV Without IFN | IVV With 10M IFN
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 29/32 | 29/32 | 26/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVV With 1M IFN (N=32) | IVV Without IFN (N=32) | IVV With 10M IFN (N=31)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 8 (8) — Solicited on the memory aid as "Cough"
Feeling hot (General disorders) | 0 (0) | 1 (1) | 2 (2) — Solicited on the memory aid as "Feverishness"
Headache (Nervous system disorders) | 14 (14) | 17 (17) | 12 (12) — Solicited on the memory aid as "Headache"
Malaise (General disorders) | 7 (7) | 11 (11) | 9 (9) — Solicited on the memory aid as "Malaise (decreased energy)"
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5) | 5 (5) — Solicited on the memory aid as "Myalgia (body aches)"
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 14 (14) | 10 (10) — Solicited on the memory aid as "Nasal discharge"
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 10 (10) | 9 (9) — Solicited on the memory aid as "Nasal obstruction"
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (6) — Solicited on the memory aid as "Nausea"
Sneezing (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 13 (13) | 9 (9) — Solicited on the memory aid as "Sneezing"
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (10) | 11 (11) — Solicited on the memory aid as "Sore throat"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less